CLINICAL TRIAL: NCT06017297
Title: Phase II Study of Neoadjuvant Durvalumab (MEDI4736) and Tremelimumab in Combination With Gemcitabine and Cisplatin in Patients With Intrahepatic Cholangiocarcinoma That is Borderline Resectable/Resectable But With High Risk for Recurrence.
Brief Title: Neoadjuvant Tremelimumab and Durvalumab With Gem/Cis in Intrahepatic Cholangiocarcinoma
Acronym: ESR-22-21719
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision and challenges in finding eligible participants
Sponsor: Georgetown University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006462
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Borderline Resectable Carcinoma; Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — durvalumab; tremelimumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Durvalumab and Tremelimumab plus gemcitabine/cisplatin (Experimental): Durvalumab and tremelimumab plus gemcitabine/cisplatin combination therapy. If the tumor is evaluated to be resectable after Cycle 4 (C4), then the patient may proceed with surgical tumor resection. If the tumor is deemed unresectable after C4, then the patient will proceed with Cycle 5-8 followed by reevaluation for surgical resection.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Gemcitabine; Drug: Cisplatin; Procedure: Surgical Resection

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500 mg via intravenous (IV) infusion every 3 weeks for up to 8 cycles
Drug: Tremelimumab — A single dose of tremelimumab at 300mg IV is given on C1.
Drug: Gemcitabine — Gemcitabine is dosed at 1000 mg/m2 IV on day (D)1 and D8 of each cycle.
Drug: Cisplatin — Cisplatin is dosed at 25mg/m2 on D1 and D8 of each cycle.
Procedure: Surgical Resection — If the tumor is evaluated to be resectable (as defined as successfully treated stage II (tumor shrink away from vessels), stage IIIA (tumor shrink away from visceral peritoneum), stage IIIB (N1 disease no longer pathologically enlarged) after C4 or C8, then the patient may proceed with surgical tumor resection.

SUMMARY:
The goal of this clinical trial is to test feasibility and safety of the combination of tremelimumab and durvalumab plus gemcitabine and cisplatin as a neoadjuvant treatment bridge patients to a curative resection in treatment naïve borderline resectable, or resectable with high risk for recurrence intrahepatic cholangiocarcinoma patients. The main question[s] it aims to answer are:

* What is the rate of conversion of unresectable tumor to resectable cancer?
* What are the side effects of this treatment combination?

Participants will undergo an initial tumor biopsy, imaging and laboratory studies prior to starting treatment with durvalumab, tremelimumab, gemcitabine and cisplatin. Participants will continue for 4 cycles and if the tumor is found to be resectable then they will undergo surgical resection. If the tumor is unresectable (can't be surgically removed) after 4 cycles, then participants will receive 4 more cycles and repeated imaging. If the tumor remains unresectable then the participant will be treated with capecitabine for up to 8 cycles and durvalumab for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age 18 years and older at the time of study entry, both sexes, all ethnicities.
2. Patients with histologically proven intrahepatic cholangiocarcinoma, untreated with systemic therapy.
3. Patients with an absence of extrahepatic metastasis (outside of periportal lymph node enlargement) or peritoneal carcinomatosis as demonstrated by CT-scan.
4. Patients with a performance status ECOG 0, 1.
5. Patients with an estimated life expectancy > 6 months.
6. Patients with disease that is not readily suitable for resection with curative intent, as validated by a multidisciplinary committee with at least one hepatobiliary surgeon, defined as stage II and stage III disease, surgical resectable if there is tumor shrinkage.
7. Patients with at least one measurable lesion according to RECIST 1.1 criteria. Tumor assessment by computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 28 days prior to start of study.
8. Patients with platelets ≥ 75,000/mm3, polynuclear neutrophils ≥ 1500/mm3, hemoglobin ≥ 9g/dL.
9. Patients with serum creatinine < 1.5 times institutional upper limit of normal (ULN), measured creatinine clearance > 40 mL/min or Calculated creatinine clearance > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24 hour urine collection for determination of creatinine clearance.
10. Patients with serum bilirubin ≤ 1.5 times institutional upper limit of normal (ULN) (after biliary drainage if necessary).
11. Absolute neutrophil count (ANC ≥ 1.0 × 109 /L)
12. Aspartate aminotransferase (AST or SGOT) / alanine transaminase (ALT or SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
13. Patients with a reference CT Scan within 30 days preceding the 1st cycle of treatment.
14. Patients with US health insurance coverage.
15. Patients are capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
16. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
17. Body weight ≥30 kg

Exclusion Criteria:

1. Patients with hilar or distal cholangiocarcinoma or those with hepatocholangiocarcinoma.
2. Patients who are eligible for surgical resection or liver transplantation based on tumor characteristics.
3. Patients who would not be surgical candidates due to reasons unrelated to their cholangiocarcinoma, e.g. Cirrhosis with portal hypertension
4. Patients with extrahepatic metastases beyond periportal lymph node enlargement
5. Patients with a contraindication or grade 3-4 allergy to durvalumab, tremelimumab, gemcitabine, cisplatin, or capecitabine.
6. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
7. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
8. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
9. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
10. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of Investigational Product (IP). Note: Local surgery of isolated lesions for palliative intent is acceptable
11. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
12. History of leptomeningeal carcinomatosis
13. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart)
14. Prior randomization or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
15. Patients with an active autoimmune disease that has required systemic treatment in the past 2 years with the use of disease-modifying agents, corticosteroids, or immunosuppressive drugs. Exceptions to this criterion include intranasal, inhaled, topical steroids or local steroid injections, systemic corticosteroids at physiologic doses not to exceed 10mg/day or prednisone or its equivalent, or steroids as premedication for hypersensitivity reactions.
16. Patients with a history of allogenic organ transplantation.
17. Patients with a history of non-infectious pneumonitis that required steroids or has current pneumonitis.
18. Patients who are recipients of a live attenuated vaccine within 30 days prior to the dose of durvalumab.
19. Patients with poorly controlled diarrhea (grade ≥ 2).
20. Coinfection of hepatitis B virus (HBV) and hepatitis C virus (HCV) as determined by viral load. HBV infection is allowed only if patient is on HBV treatment per institutional guideline. HCV infection is allowed.
21. Patients known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice)
22. Patients with a serious, non-stabilized disease, active uncontrolled infection, or other serious underlying disorders that would likely prevent the patient from receiving therapy.
23. Patients who are pregnant, breast-feeding, or of child-bearing age with a refusal to use effective contraception.
24. Patients with another cancer, active within the 5 years preceding or at the time of inclusion in this trial. Note: Patients with early-stage cancer that has been resected/ablated/radiated, without evidence of disease recurrence or progression, within 2 years may be considered.
25. Patients with legal incapacity.
26. Patients who are deprived of civil liberty.
27. Patients for whom it is impossible to sign the informed consent document or to adhere to medical follow-up of the trial for geographical, social, or psychological reasons.
28. Patients who have participation in another clinical study with an investigational product during the last 4 weeks.
29. Patients who are concurrently enrolled in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
30. Patients who are judged by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with the study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Rate of Conversion from unresectable to resectable | 8 Cycles, 21 day cycles
  Rate of conversion of unresectable tumor to resectable cancer after neoadjuvant durvalumab + tremelimumab + gemcitabine + cisplatin after 4 or 8 cycles. Surgical evaluation will be done in joint by institutional radiology and hepatobiliary surgery using clinical data (CT/MRI imaging, patient performance status, labs, etc.) If among the evaluable 24 patients, 9 or more (45%) patients undergo such conversion, the investigational treatment will be considered as promising/feasible. The resectable rate will be estimated with its 95% exact confidence interval.
Incidence of related treatment emergent adverse events | 36 months
  Number of participants with related treatment emergent adverse events

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 36 months
  ORR will be estimated with its 95% exact confidence interval based on RECIST v1.1
Pathological complete response (pCR) | 36 months
Overall survival (OS) | 36 months
  Kaplan-Meier method is used to represent secondary outcome OS.
Progression-free survival (PFS) | 36 months
  Kaplan-Meier method is used to represent secondary outcome of PFS
Rate of R0 resection | 8 Cycles, 21 day cycles
  R0 resection rate will be estimated with its 95% exact confidence interval
Relapse free survival (RFS) | 36 months
  Kaplan-Meier method will be used to analyze RFS
Patient Reported outcomes (PRO) decline | 8 Cycles, 21 day cycles
  As measured by qualify of life changes per EORTC QLQ-BIL-20 questionnaires. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Event Free Survival (EFS) | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Aiwu R He, MD, Principal Investigator — Georgetown University

IPD SHARING:
Plan to Share IPD: No